CLINICAL TRIAL: NCT04134091
Title: A Phase 2, Randomized Double-Blind, Placebo-Controlled, Multi-Center Study to Assess the Efficacy, Safety and Tolerability of Oral LPCN 1144 in Subjects With Nonalcoholic Steatohepatitis (NASH)
Brief Title: The Efficacy, Safety and Tolerability of Oral LPCN 1144 in Subjects With Nonalcoholic Steatohepatitis
Acronym: NASH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lipocine Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LPCN 1144-18-002
Record Dates: First submitted 2019-08-16; First posted 2019-10-21 (Actual); Results first posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Nonalcoholic Steatohepatitis (NASH)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — testosterone undecanoate; alpha-Tocopherol

STUDY DESIGN:
Intervention Model Description: Randomized in 1:1:1 ratio to receive one of the following treatments:
  * Treatment A: Oral LPCN 1144 Formulation A
  * Treatment B: Oral LPCN 1144 Formulation B
  * Treatment C: Oral matching placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects meeting the enrollment criteria will be randomly assigned to one of the three treatment arms. The randomization will be carried out by central assignment. The study is a blinded study; therefore all the randomization codes will be centrally maintained and no data from the randomization will be available to Sponsor, contract research organization (CRO) operations team, medical monitors, monitors or any site staff.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment A (Experimental): LPCN 1144 Formulation A
  Interventions: Drug: LPCN 1144 Formulation A
- Treatment B (Experimental): LPCN 1144 Formulation B
  Interventions: Drug: LPCN 1144 Formulation B
- Treatment C (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LPCN 1144 Formulation A — Oral LPCN 1144 Formulation A capsule, total daily dose of 450 mg testosterone undecanoate administered as 225 mg testosterone undecanoate twice daily (BID).
  Other Names: testosterone undecanoate
  Arms: Treatment A
Drug: LPCN 1144 Formulation B — Oral LPCN 1144 + d-alpha tocopherol total daily dose of 450 mg testosterone undecanoate + 476 mg d-alpha tocopherol administered as 225 mg testosterone undecanoate + 238 mg d-alpha tocopherol BID
  Other Names: testosterone undecanoate with d-alpha tocopherol
  Arms: Treatment B
Drug: Placebo — Oral matching placebo capsule administered as BID
  Other Names: Oral placebo
  Arms: Treatment C

SUMMARY:
This is a Phase 2, randomized, double-blind, placebo controlled, three arm study in adult men with biopsy confirmed NASH. The study is aimed at evaluating efficacy and tolerability of LPCN 1144 in adult men with NASH.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-blind, placebo controlled, three arm study in adult men with biopsy confirmed NASH. The study is aimed at evaluating efficacy and tolerability of LPCN 1144 in adult men with NASH. The study will be conducted across multiple centers in the United States.

Approximately 75 subjects will be randomized in 1:1:1 ratio to receive one of the following treatments:

* Treatment A: Oral LPCN 1144 Formulation A
* Treatment B: Oral LPCN 1144 Formulation B
* Treatment C: Oral matching placebo

Subjects will undergo a screening period to determine study eligibility. As a part of screening, liver biopsies will be performed for subjects who have not had a liver biopsy within 6 months of Day 1, and fat fraction will be measured by magnetic resonance imaging derived proton density fat fraction (MRI-PDFF) in all subjects. Adult male subjects with histologic evidence of NASH will be enrolled into the study.

Eligible subjects will be randomized to one of the three treatment arms. The treatment phase will be for a duration of 36-weeks with assessments of liver biopsies, hepatic fat fraction, liver enzymes, lipid levels and other safety parameters. Safety and tolerability will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male between 18 and 80 years of age, inclusive.
2. Subject with histologic evidence of NASH upon central read of a liver biopsy.

   i. A historical biopsy no more than 4 months before Screening may be considered for use with medical monitor approval if the following criteria are met:
   * Stable weights between the time of the biopsy and Screening. Stable weight is defined as no more than a 5% change.
   * Is either not taking or is on a stable dose of Thiazolidinedione(TZDs)/glitazones for 3 months before Day 1.
3. Background therapy for other ongoing chronic conditions, and weight should be stable for at least 3 months before trial enrollment. Stable weight is defined as no more than a 5% change.
4. Judged to be in good general health as determined by the investigator at screening.

Exclusion Criteria:

1. Significant alcohol consumption more than 30 g/day on average, either currently or for a period of more than 3 consecutive months in the 5 years prior to screening.
2. Inability to reliably quantify alcohol intake.
3. Biochemical, clinical or histologic evidence of cirrhosis on liver biopsy (stage 4 fibrosis).
4. Evidence of other causes of chronic liver disease including alcoholic liver disease, viral hepatitis, primary biliary cirrhosis, primary sclerosing cholangitis, autoimmune hepatitis, Wilson's disease, hemochromatosis, alpha-1 antitrypsin deficiency, human immunodeficiency virus, etc.
5. Suspected or proven liver cancer.
6. Clinically significant abnormal laboratory value, in the opinion of the investigator, in serum chemistry, hematology, or urinalysis including but not limited to:

   * Hematocrit > upper limits of normal (ULN)
   * Hemoglobin > ULN
   * Prostate-specific antigen (PSA) > 4 ng/mL
   * Serum aspartate aminotransferase (AST) or alanine transaminase (ALT) > 200 IU/L
   * Serum alkaline phosphatase (ALP) > 2 x ULN
   * Serum creatinine of 2.0 mg/dL or greater
   * Total bilirubin > ULN
   * International normalized ratio (INR) ≥ 1.3.
   * Prolactin > ULN
7. Subjects with evidence of worsening liver function based on the two initial laboratory values used to establish the screening / baseline values.
8. Model for End-Stage Liver Disease (MELD) score greater than 12
9. Subjects with a documented history of Gilbert's syndrome
10. Evidence of portal hypertension (e.g., low platelet counts, esophageal varices, ascites, history of hepatic encephalopathy, splenomegaly).
11. Use of drugs historically associated with NAFLD (amiodarone, methotrexate, systemic glucocorticoids, tetracyclines, tamoxifen, estrogens, anabolic steroids, valproic acid, other known hepatotoxins) for more than 2 weeks in the 2 years prior to randomization.
12. Subjects who are not on a stable dose of lipid-lowering drugs, diabetic and / or hypertensive medication in the 3 months prior to biopsy or the 3 months prior to randomization
13. Any over-the-counter medication or herbal remedy that is being taken with an intent to improve hyperlipidemia must be stable for at least 3 months prior to randomization and through the end of the study.
14. Vitamin E supplementation of greater than 100 IU/day, unless completed adequate washout for at least 4 weeks prior to Day 1 or biopsy if one is required.
15. Inability to safely obtain a liver biopsy.
16. History of total parenteral nutrition in the year prior to screening.
17. History of bariatric surgery or currently undergoing evaluation for bariatric surgery.
18. History of gastric surgery, vagotomy, bowel resection or any surgical procedure that might interfere with gastrointestinal motility, pH or absorption.
19. History of biliary diversion.
20. Known positivity for antibody to Human Immunodeficiency Virus (HIV).
21. Known heart failure of New York Heart Association class 3 or 4.
22. Active, serious medical disease with likely life-expectancy less than 5 years.
23. History of current or suspected prostate or breast cancer.
24. History of diagnosed, severe, untreated, obstructive sleep apnea.
25. Active substance abuse in the year prior to screening.
26. History of significant sensitivity or allergy to any androgens, including testosterone, or product excipients
27. History of seizures or convulsions, including alcohol or drug withdrawal seizures. Childhood seizures are not exclusionary.
28. Use of known strong inhibitors (e.g., ketoconazole) or inducers (e.g., dexamethasone, phenytoin, rifampin, carbamazepine) of cytochrome P450 3A (CYP3A) within 30 days prior to study drug administration and through the end of the study.
29. Subjects who are currently receiving any androgens (testosterone or other androgens or androgen supplements). Subjects who are on testosterone may be eligible for the study following an adequate washout (12 weeks following intramuscular androgen injections; 4 weeks following topical or buccal androgens; 3 weeks following oral androgens).
30. Use of any investigational drug within 5 half-lives of the last dose or in the past 6 months prior to Study Day -2 without PI and/or Sponsor approval.
31. Receipt of any drug by injection within 30 days or 10 half-lives (whichever is longer) prior to study drug administration without PI and/or Sponsor approval. Insulin, allergy shots, and vaccines are allowed.
32. Subject who is not willing to use adequate contraception for the duration of the study.
33. Any other condition, which in the opinion of the investigator would impede compliance or hinder completion of the study.
34. Failure to give informed consent.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony DelConte, Study Director — Lipocine Inc.
Locations (19):
- United States (19):
  - TriWest Research Associates, LLC, El Cajon, California
  - United Medical Doctors, Murrieta, California
  - Inland Empire Liver Foundation, Rialto, California
  - Clinical Trials Research, Roseville, California
  - Meridien Research-Maitland, Maitland, Florida
  - Clinical Pharmacology of Miami, LLC, Miami, Florida
  - Sensible Healthcare, LLC, Ocoee, Florida
  - Tandem Clinical Research, Marrero, Louisiana
  - Jubilee Clinical Research, Inc., Las Vegas, Nevada
  - Clinical Research of South Nevada, Las Vegas, Nevada
  - Awasty Research Network, Marion, Ohio
  - R&H Clinical Research, Katy, Texas
  - Sun Research Institute, San Antonio, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - Clinical Trial Network-Houston, Spring, Texas
  - Pioneer Research Soultions, Sugar Land, Texas
  - Advanced Clinical Research - Gut Whisperer, Riverton, Utah
  - Granger Medical Clinic, West Valley City, Utah
  - Manassas Clinical Research Center, Manassas, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment A: LPCN 1144 Formulation A
  LPCN 1144 Formulation A: Oral LPCN 1144 Formulation A capsule, total daily dose of 450 mg testosterone undecanoate administered as BID (225 mg testosterone undecanoate per dose)
- Treatment B: LPCN 1144 Formulation B
  LPCN 1144 Formulation B: Oral LPCN 1144 + d-alpha tocopherol total daily dose of 450 mg testosterone undecanoate + 476 mg d-alpha tocopherol administered as BID (225 mg testosterone undecanoate + 238 mg d-alpha tocopherol per dose)
Period: Overall Study
Arm/Group | Treatment A | Treatment B | Treatment C
Started | 18 | 19 | 19
Completed Week 12 | 18 | 19 | 18
Completed | 18 (Completed Week 36) | 17 (Completed Week 36) | 17 (Completed Week 36)
Not Completed | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment A | Treatment B | Treatment C | Total
Number analyzed (Participants) | 18 | 19 | 19 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 15 | 15 | 47
  >=65 years | 1 | 4 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (8.66) | 53.4 (10.68) | 53.6 (11.2) | 52.8 (10.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 18 | 19 | 19 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 6 | 19
  Not Hispanic or Latino | 11 | 13 | 13 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2
  White | 18 | 18 | 16 | 52
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Hepatic Fat Fraction Based on MRI-PDFF Measurements in LPCN 1144 Treated Subjects Compared to Placebo.
Description: The change in magnetic resonance imaging derived proton fat fraction (MRI-PDFF) from baseline to week 12 in LPCN 1144 treated subjects and subjects given placebo.
Time Frame: Baseline and Week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of liver fat
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 18 | 19 | 19
Percentage of liver fat | -7.68 [-9.82 to -5.54] | -9.17 [-11.26 to -7.08] | -1.54 [-3.65 to 0.58]
Statistical Analysis 1: Comparison: Treatment A vs Treatment C; Test type: Superiority; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Treatment B vs Treatment C; Test type: Superiority; p < 0.0001, ANCOVA

2. Secondary Outcome: Relative Change in MRI-PDFF Measurements in LPCN 1144 Treated Subjects Compared to Placebo.
Description: Requirement for inclusion in analysis was having a baseline hepatic fat fraction ≥ 5% based on MRI-PDFF.
Time Frame: Baseline and week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 17 | 17 | 18
Percentage change | -39.94 [-50.76 to -29.11] | -46.84 [-57.30 to -36.38] | -9.34 [-20.20 to 1.53]
Statistical Analysis 1: Comparison: Treatment A vs Treatment C; Test type: Superiority; p = 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Treatment B vs Treatment C; Test type: Superiority; p < 0.0001, ANCOVA

3. Secondary Outcome: Number of Participants With Resolution of NASH on Overall Histopathological Reading in LPCN 1144 Treated Subjects Compared to Placebo
Description: Resolution of nonalcoholic steatohepatitis (NASH) is defined as the nonalcoholic fatty liver disease activity score (NAS) score of 0-1 for inflammation, 0 for ballooning, and any value for steatosis. These data are based on the NASH-clinical research network (CRN) histology scoring system. The range of scores are as follows (with higher scores equating to a more pathological feature): Steatosis 0-3, inflammation 0-3, ballooning 0-2, fibrosis state 0-4, and NAS 0-8.
Time Frame: Baseline and Week 36
Population: Number of participants reflect the participants who had NASH at baseline, as confirmed by a biopsy, and a second biopsy at week 36.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 13 | 13 | 11
Participants | 7 | 9 | 1
Statistical Analysis 1: Comparison: Treatment A vs Treatment C; Test type: Superiority; p < 0.05, Fisher Exact
Statistical Analysis 2: Comparison: Treatment B vs Treatment C; Test type: Superiority; p < 0.01, Fisher Exact

4. Secondary Outcome: Number of Subjects Achieving Resolution of NASH on Overall Histopathological Reading and no Worsening of Liver Fibrosis in LPCN 1144 Treated Subjects Compared to Placebo.
Description: Resolution of NASH is defined as NAS score of 0-1 for inflammation, 0 for ballooning, and any value for steatosis. These data are based on the NASH-CRN histology scoring system. The range of scores are as follows (with higher scores equating to a more pathological feature): Steatosis 0-3, inflammation 0-3, ballooning 0-2, fibrosis state 0-4, and NAS 0-8. No worsening was defined as a score in fibrosis equal to, or lower, than baseline.
Time Frame: Baseline and Week 36
Population: Overall number of participants reflect the participants who had NASH at baseline, as confirmed by a biopsy, and a second biopsy at week 36.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 13 | 13 | 11
Participants | 6 | 9 | 0
Statistical Analysis 1: Comparison: Treatment A vs Treatment C; Test type: Superiority; p < 0.05, Fisher Exact
Statistical Analysis 2: Comparison: Treatment B vs Treatment C; Test type: Superiority; p < 0.001, Fisher Exact

5. Secondary Outcome: Number of Subjects With Improvement in NASH Evaluated by Paired Biopsies Analysis and no Worsening of Liver Fibrosis in LPCN 1144 Treated Subjects Compared to Placebo.
Description: Paired biopsies are randomly assigned A or B and are scored by a blinded pathologist as better, worse or same for change in fibrosis, steatosis, inflammation, and ballooning. Improvement in NASH requires no worsening of fibrosis, an improvement in ballooning or inflammation, and no worsening of ballooning or inflammation. Assessment of better or same is considered as no worsening.
Time Frame: Baseline and week 36
Population: Overall number of participants are based on those with a baseline and week 36 biopsy
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 15 | 14 | 15
Participants | 9 | 8 | 2
Statistical Analysis 1: Comparison: Treatment A vs Treatment C; Test type: Superiority; p < 0.05, Fisher Exact
Statistical Analysis 2: Comparison: Treatment B vs Treatment C; Test type: Superiority; p < 0.05, Fisher Exact

6. Secondary Outcome: Change in the Mean Score of NAS Components at Baseline and After 36 Weeks of Treatment in LPCN 1144 Treated Subjects Compared to Placebo.
Description: These data are based on the NASH-CRN histology scoring system. The range of scores are as follows (with higher scores equating to a more pathological feature): Steatosis 0-3, inflammation 0-3, ballooning 0-2, fibrosis state 0-4, and NAS 0-8.
Time Frame: Baseline and Week 36
Population: Overall number of participants are based on those with a baseline and week 36 biopsy.
Measure: Least Squares Mean (95% Confidence Interval); unit: NAS score
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 15 | 14 | 15
NAS score
  Hepatocyte ballooning score | -0.7 [-1.1 to -0.3] | -0.9 [-1.3 to -0.5] | -0.2 [-0.6 to 0.2]
  Lobular inflammation score | -0.2 [-0.5 to 0.1] | -0.5 [-0.8 to -0.1] | -0.1 [-0.4 to 0.2]
  Steatosis score | -0.9 [-1.3 to -0.6] | -1.2 [-1.6 to -0.8] | -0.1 [-0.5 to 0.2]
Statistical Analysis 1: Comparison: Treatment A vs Treatment C; Outcome Variable: Hepatocyte Ballooning Score; Test type: Superiority; p > 0.05, ANCOVA
Statistical Analysis 2: Comparison: Treatment B vs Treatment C; Outcome Variable: Hepatocyte Ballooning Score; Test type: Superiority; p < 0.05, ANCOVA
Statistical Analysis 3: Comparison: Treatment A vs Treatment C; Outcome Variable: Lobular Inflammation Score; Test type: Superiority; p > 0.05, ANCOVA
Statistical Analysis 4: Comparison: Treatment B vs Treatment C; Outcome Variable: Lobular Inflammation Score; Test type: Superiority; p > 0.05, ANCOVA
Statistical Analysis 5: Comparison: Treatment A vs Treatment C; Outcome Variable: Steatosis Score; Test type: Superiority; p < 0.01, ANCOVA
Statistical Analysis 6: Comparison: Treatment B vs Treatment C; Outcome Variable: Steatosis Score; Test type: Superiority; p < 0.001, ANCOVA

7. Secondary Outcome: Number of Subjects With an Improvement in Liver Fibrosis Greater Than or Equal to One Stage and no Worsening of NASH in LPCN 1144 Treated Subjects Compared to Placebo.
Description: These data are based on the NASH-CRN histology scoring system. The range of scores are as follows (with higher scores equating to a more pathological feature): Steatosis 0-3, inflammation 0-3, ballooning 0-2, and fibrosis stage 0-4. Improvement in liver fibrosis was defined as an improvement in fibrosis greater than or equal to one stage using the NASH CRN fibrosis score with no worsening of ballooning, inflammation, or steatosis.
Time Frame: Baseline and Week 36
Population: Overall number of participants are based on those with a baseline and week 36 biopsy.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 15 | 14 | 15
Participants | 4 | 2 | 6
Statistical Analysis 1: Comparison: Treatment A vs Treatment C; Test type: Superiority; p > 0.05, Fisher Exact
Statistical Analysis 2: Comparison: Treatment B vs Treatment C; Test type: Superiority; p > 0.05, Fisher Exact

8. Secondary Outcome: Number of Subjects With Improvement in Fibrosis Evaluated by Paired Biopsies Analysis and no Worsening of NASH in LPCN 1144 Treated Subjects Compared to Placebo
Description: Paired biopsies are randomly assigned A or B and are scored by a blinded pathologist as better, worse or same for change in fibrosis, steatosis, inflammation, and ballooning. Improvement in fibrosis requires a better score in fibrosis and no worsening of ballooning or inflammation. Assessment of better or same is considered as no worsening.
Time Frame: Baseline to week 36
Population: Overall number of participants are based on those with a baseline and week 36 biopsy.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 15 | 14 | 15
Participants | 6 | 8 | 3
Statistical Analysis 1: Comparison: Treatment A vs Treatment C; Test type: Superiority; p > 0.05, Fisher Exact
Statistical Analysis 2: Comparison: Treatment B vs Treatment C; Test type: Superiority; p > 0.05, Fisher Exact

9. Secondary Outcome: Number of Subjects With Improvement in Fibrosis Evaluated Via FibroNest Scores
Description: Improvement in Fibrosis is defined as improvement in parenchymal tissue normalized phenotypic fibrosis composite value compared to baseline. FibroNest is an image analysis system for the assessment of the severity and progression of fibrosis in NASH, produced by PharmaNest LLC.
Time Frame: Baseline and week 36
Population: Overall number of participants are based on those with a baseline and week 36 biopsy.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 15 | 14 | 15
Participants | 12 | 6 | 5
Statistical Analysis 1: Comparison: Treatment A vs Treatment C; Test type: Superiority; p < 0.05, Fisher Exact
Statistical Analysis 2: Comparison: Treatment B vs Treatment C; Test type: Superiority; p > 0.05, Fisher Exact

10. Secondary Outcome: Relative Change in Appendicular Lean Muscle Mass
Description: Relative change in appendicular lean muscle mass measured by dual-energy absorptiometry (DXA) in LPCN 1144 treated subjects compared to Placebo. Data were last observation carried forward.
Time Frame: Baseline and 36 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 13 | 13 | 14
Percentage change | 2.75 [-0.04 to 5.54] | 1.90 [-0.87 to 4.67] | -1.42 [-4.12 to 1.28]
Statistical Analysis 1: Comparison: Treatment A vs Treatment C; Test type: Superiority; p < 0.05, ANCOVA
Statistical Analysis 2: Comparison: Treatment B vs Treatment C; Test type: Superiority; p > 0.05, ANCOVA

11. Secondary Outcome: Relative Change in Whole Body Fat Mass
Description: Relative change in whole body fat mass measured by dual-energy absorptiometry (DXA) in LPCN 1144 treated subjects compared to Placebo. Data were last observation carried forward.
Time Frame: Baseline and week 36
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 13 | 13 | 14
Percentage change | -3.68 [-9.60 to 2.24] | -7.33 [-13.35 to -1.31] | 1.78 [-4.01 to 7.57]
Statistical Analysis 1: Comparison: Treatment A vs Treatment C; Test type: Superiority; p > 0.05, ANCOVA
Statistical Analysis 2: Comparison: Treatment B vs Treatment C; Test type: Superiority; p < 0.05, ANCOVA

12. Secondary Outcome: Mean Change From Baseline in Liver Enzymes in LPCN 1144 Treated Subjects Compared to Placebo.
Description: Liver enzymes analyzed were aspartate transaminase (AST), alanine transaminase (ALT), alkaline phosphatase (ALP), and gamma-glutamyltransferase (GGT)
Time Frame: Baseline and Week 36
Measure: Least Squares Mean (95% Confidence Interval); unit: U/L
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 18 | 17 | 17
U/L
  Aspartate transaminase (AST) | -8.0 [-14.9 to -1.0] | -12.0 [-18.9 to -5.1] | 1.3 [-5.8 to 8.3]
  Alanine transaminase (ALT) | -11.4 [-23.1 to 0.3] | -22.9 [-34.5 to -11.2] | 0.6 [-11.3 to 12.4]
  Alkaline phosphatase (ALP) | -6.1 [-11.4 to -0.9] | -8.5 [-13.7 to -3.3] | 0.1 [-5.1 to 5.4]
  Gamma-glutamyltransferase (GGT) | -2.9 [-11.4 to 5.6] | -13.4 [-22.0 to -4.9] | 0.7 [-8.0 to 9.4]
Statistical Analysis 1: Comparison: Treatment A vs Treatment C; Outcome Variable: AST; Test type: Superiority; p > 0.05, Mixed Models Analysis
Statistical Analysis 2: Comparison: Treatment B vs Treatment C; Outcome Variable: AST; Test type: Superiority; p < 0.01, Mixed Models Analysis
Statistical Analysis 3: Comparison: Treatment A vs Treatment C; Outcome Variable: ALT; Test type: Superiority; p > 0.05, Mixed Models Analysis
Statistical Analysis 4: Comparison: Treatment B vs Treatment C; Outcome Variable: ALT; Test type: Superiority; p < 0.01, Mixed Models Analysis
Statistical Analysis 5: Comparison: Treatment A vs Treatment C; Outcome Variable: ALP; Test type: Superiority; p > 0.05, Mixed Models Analysis
Statistical Analysis 6: Comparison: Treatment B vs Treatment C; Outcome Variable: ALP; Test type: Superiority; p < 0.05, Mixed Models Analysis
Statistical Analysis 7: Comparison: Treatment A vs Treatment C; Outcome Variable: GGT; Test type: Superiority; p > 0.05, Mixed Models Analysis
Statistical Analysis 8: Comparison: Treatment B vs Treatment C; Outcome Variable: GGT; Test type: Superiority; p < 0.05, Mixed Models Analysis

13. Secondary Outcome: Mean Changes in Serum Lipid Profile Parameters in LPCN 1144 Treated Subjects Compared to Placebo.
Description: Lipid profile parameters included total cholesterol, low-density lipoprotein (LDL), high-density lipoprotein (HDL), and triglycerides.
Time Frame: Baseline and Week 36
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 18 | 17 | 16
mg/dL
  Total Cholesterol | -1.7 [-17.7 to 14.2] | 7.3 [-8.8 to 23.4] | 1.1 [-15.4 to 17.7]
  LDL | 1.8 [-11.4 to 15.1] | 8.7 [-3.6 to 21.1] | -6.0 [-20.0 to 7.9]
  HDL | -3.3 [-5.8 to -0.7] | -2.0 [-4.6 to 0.6] | -0.0 [-2.7 to 2.7]
  Triglycerides | -11.5 [-78.6 to 55.6] | -3.9 [-70.8 to 63.0] | 67.3 [-0.2 to 134.9]
Statistical Analysis 1: Comparison: Treatment A vs Treatment C; Outcome Variable: Total cholesterol; Test type: Superiority; p > 0.05, Mixed Models Analysis
Statistical Analysis 2: Comparison: Treatment B vs Treatment C; Outcome Variable: Total cholesterol; Test type: Superiority; p > 0.05, Mixed Models Analysis
Statistical Analysis 3: Comparison: Treatment A vs Treatment C; Outcome Variable: LDL; Test type: Superiority; p > 0.05, Mixed Models Analysis
Statistical Analysis 4: Comparison: Treatment B vs Treatment C; Outcome Variable: LDL; Test type: Superiority; p > 0.05, Mixed Models Analysis
Statistical Analysis 5: Comparison: Treatment A vs Treatment C; Outcome Variable: HDL; Test type: Superiority; p > 0.05, Mixed Models Analysis
Statistical Analysis 6: Comparison: Treatment B vs Treatment C; Outcome Variable: HDL; Test type: Superiority; p > 0.05, Mixed Models Analysis
Statistical Analysis 7: Comparison: Treatment A vs Treatment C; Outcome Variable: triglycerides; Test type: Superiority; p > 0.05, Mixed Models Analysis
Statistical Analysis 8: Comparison: Treatment B vs Treatment C; Outcome Variable: triglycerides; Test type: Superiority; p > 0.05, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for a duration of 36 weeks for each participant while enrolled in study.
Arm/Group | Treatment A | Treatment B | Treatment C
All-Cause Mortality (participants affected / at risk) | 1/18 | 0/19 | 1/19
Serious Adverse Events (participants affected / at risk) | 2/18 | 2/19 | 1/19
Other Adverse Events (participants affected / at risk) | 12/18 | 11/19 | 16/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=18) | Treatment B (N=19) | Treatment C (N=19)
Corona virus infection (Infections and infestations) | 0 | 1 | 1
Polycythemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Hyperprolactinemia (Endocrine disorders) | 1 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Mental status change (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=18) | Treatment B (N=19) | Treatment C (N=19)
Corona virus infection (Infections and infestations) | 2 | 1 | 2
Bronchitis (Infections and infestations) | 1 | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 2 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Latent tuberculosis (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0 | 0
Oral muscosal blistering (Gastrointestinal disorders) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1
Coronavirus test postive (Investigations) | 1 | 0 | 0
Cortisol decreased (Investigations) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0
Glycosylated hemoglobin increased (Investigations) | 0 | 0 | 1
Hematocrit increased (Investigations) | 0 | 1 | 0
Prostatic specific antigen increased (Investigations) | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 2
Hypercholesterolemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperlipidemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 3 | 0 | 1
Aortic arteriosclerosis (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0
Edema peripheral (General disorders) | 1 | 1 | 2
Pyrexia (General disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 1
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 1 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus generalized (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash generalized (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Retinal tear (Eye disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Hyperprolactinemia (Endocrine disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT04134091/Prot_002.pdf
  • Statistical Analysis Plan (2021-03-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT04134091/SAP_003.pdf